CLINICAL TRIAL: NCT00822666
Title: Effect of the Genetic Variant 2C19*2 on Clopidogrel Biological Response in Patients With Premature Coronary Artery Disease
Brief Title: Clopidogrel and Response Variability Investigation Study 2
Acronym: CLOVIS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P070117
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Artery Disease
Keywords: Platelet aggregation; Platelet; Thrombosis; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): patients homozygous for the 2C19*1 genetic variant
  Interventions: Drug: clopidogrel
- 2 (Experimental): carriers of the 2C19*2 genetic variant (homozygous or heterozygous)
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — comparison of two loading strategies of clopidogrel (300mg vs 900mg) in the two genetic profiles

SUMMARY:
To evaluate the role of the genetic variant 2C19*2 on the pharmacodynamic response as assessed by optical aggregometry and on the pharmacokinetic response as assessed by measuring active metabolites following an oral administration of a loading dose of 300/900mg of clopidogrel in patients with established coronary artery disease.

DETAILED DESCRIPTION:
Rationale : Clopidogrel is a specific and irreversible of the P2Y12 platelet receptor leading to an inhibition of platelet aggregation. Clopidogrel is a prodrug that must be converted into an active metabolite that selectively and irreversibly binds to the P2Y12 platelet membrane receptor. As a consequence, a loading dose of 300 mg is necessary in percutaneous coronary intervention and in acute coronary syndrome, situations which require a rapid inhibition of platelet aggregation due to the high thrombotic risk.

High platelet reactivity on clopidogrel may be due to various reasons including polymorphism in the gene encoding the cytochrome P-450 2C19 enzyme (CYP2C19) which has been shown to contribute to the variability of platelet response to clopidogrel. CYP2C19 is a key enzyme in this activation process and our group was the first to describe an association between the presence of the loss of function CYP2C19 681G>A polymorphism (also called *2) with lower clopidogrel responsiveness in healthy subjects.

Poor responsiveness to clopidogrel has become a major concern given acute recurrent events following stent placement.

Objective : To evaluate the role of the genetic variant 2C19*2 on the pharmacodynamic response as assessed by optical aggregometry and on the pharmacokinetic response as assessed by measuring active metabolites following an oral administration of a loading dose of 300/900mg of clopidogrel in patients with established coronary artery disease.

Target population :Patients of less than 45 years of age and who survived a MI and enrolled in the AFIJI multicenter registry (Appraisal of risk Factors in young Ischemic patients Justifying aggressive Intervention).

Primary end-point :Comparison of inhibition of the intensity of residual platelet aggregation (IRPA) measured 6 minutes after induction by 20 μmol/L following 300mg or 900 mg of clopidogrel with respect to the presence of the genetic variant CYP2C19*2

1. Maximum platelet aggregation instead of IRPA
2. RPA with 5µM and 50 µM of ADP
3. Measure of clopidogrel and its active metabolites (carboxylated and thiol) at different time points following the loading dose (H0, H1, H2 et H6) with respect to the presence of the genetic variant CYP2C19*2
4. Relationship between active metabolites concentration and IRPA
5. Relationship between active metabolites and dose of clopidogrel
6. Comparison of 300mg vs 900mg on IRPA in the whole population irrespective of the genetic variant

Statistical analysis :Comparison of IRPA with respect to the presence of the genetic variant 2C19*2 by anova Area under the curve of the production of active metabolites with respect to the presence of the genetic variant 2C19*2 Agenda :November 2008 (inclusion of first patient) to december 2009 (analysis of the data)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Male gender
* Included in the AFIJI registry
* No high bleeding risk profile
* No recent history of acute coronary syndrome (< 3 months)
* Written informed consent obtained
* Genotype CYP2C19 : *1/*1, *1/*2 ou *2/*2
* Genotype P2Y12 : H1/H1 ou H1/H2

Exclusion Criteria:

* Female gender
* Patient with a contraindication to clopidogrel
* Patient who has received a loading dose of clopidogrel in the past 7 days
* Patient treated with ticlopidine or GP2B/3A receptor antagonist prior to loading
* Non compliance
* Génotype P2Y12 : H2/H2.
* Patient treated with drugs interacting with platelet aggregation (NSAID, persantine, serotonin inhibitors )
* Patient treated with drugs interacting 2C19
* Not affiliated to the national health insurance
* Patient participating to another randomized study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Inhibition of residual platelet activity 6 hours after a loading dose of clopidogrel | 6 hours

SECONDARY OUTCOMES:
Maximum platelet aggregation instead of IRPA | during the study
RPA with 5µM and 50 µM of ADP | during the study
3. Measure of clopidogrel and its active metabolites (carboxylated and thiol) at different time points following the loading dose (H0, H1, H2 ,H6) with respect to the presence of the genetic variant CYP2C19*2 | H0, H1, H2, H6
Relationship between active metabolites concentration and IRPA | during the study
Relationship between active metabolites and dose of clopidogrel | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Collet, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital la Pitié-Salpétrière Institut de cardiologie, Paris, France

REFERENCES:
- [Derived] Hulot JS, Collet JP, Cayla G, Silvain J, Allanic F, Bellemain-Appaix A, Scott SA, Montalescot G. CYP2C19 but not PON1 genetic variants influence clopidogrel pharmacokinetics, pharmacodynamics, and clinical efficacy in post-myocardial infarction patients. Circ Cardiovasc Interv. 2011 Oct 1;4(5):422-8. doi: 10.1161/CIRCINTERVENTIONS.111.963025. Epub 2011 Oct 4. PMID 21972404
- [Derived] Collet JP, Hulot JS, Anzaha G, Pena A, Chastre T, Caron C, Silvain J, Cayla G, Bellemain-Appaix A, Vignalou JB, Galier S, Barthelemy O, Beygui F, Gallois V, Montalescot G; CLOVIS-2 Investigators. High doses of clopidogrel to overcome genetic resistance: the randomized crossover CLOVIS-2 (Clopidogrel and Response Variability Investigation Study 2). JACC Cardiovasc Interv. 2011 Apr;4(4):392-402. doi: 10.1016/j.jcin.2011.03.002. PMID 21511218